CLINICAL TRIAL: NCT05883345
Title: Validation of Blood Test Finding for the Diagnosis of Gastritis and Gastric Neoplasms
Brief Title: Blood Tests for Gastritis and Gastric Neoplasms
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-04-056
Record Dates: First submitted 2023-05-09; First posted 2023-05-31 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Cancer Screening Tests
Keywords: Helicobacter pylori; Atrophic gastritis; Gastric cancer; Pepsinogen
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum blood test for Helicobacter pylori immunoglobulin G, pepsinogen, and gastrin-17 levels — Endoscopic biopsy
  Other Names: Upper gastrointestinal endoscopy; Urea breath test

SUMMARY:
Helicobacter pylori infection rate is decreasing in younger population; however, biennial gastroscopy is still recommended for all Koreans aged between 40 and 75 years. This study aimed to validate blood tests for gastric cancer screening according to the infection status of H. pylori (naive, current, and past infection).

DETAILED DESCRIPTION:
Helicobacter pylori-seropositive rates are decreasing in South Korea. Seroprevalence was 74.3% in 1990, but it decreased to 43.9% in 2016. In Koreans, most gastric cancers are related to H. pylori infection. H. pylori-negative gastric cancers were found only in 2.3% among the 1,833 Korean gastric cancer patients. Despite these facts, the national guideline still recommends biennial gastroscopy for all Koreans aged between 40 and 75 years. Therefore, 8,462,570 (63.1%) Koreans underwent gastric cancer screening among the target population of 13,404,927 individuals in 2021.

In H. pylori-seroprevalent populations, diagnostic criteria for naive status should be strict based on histology, endoscopy, and serum pepsinogen (PG) assay findings. Naive condition should be diagnosed only when both invasive and non-invasive H. pylori tests show negative findings. Furthermore, there should be no intestinal metaplasia and atrophy on serum PG assay, endoscopy, and histology findings in H. pylori-naive participants. Based on those findings, H. pylori infection will be confirmed when invasive tests or urea breath test was positive. H. pylori-naive status will be diagnosed if there was no eradication history, no serologically detected atrophy (PG I ≤70 ng/mL and PG I/II ≤3), and no intestinal metaplasia or atrophy on endoscopy and histology.

This study aimed to determine the validity of blood tests for gastric cancer screening according to the H. pylori infection status. We tried to identify significant variables using GastroPanel tests and traditional serum PG assays in patients with gastric neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who visited for gastric cancer screening

Exclusion Criteria:

* History of gastrectomy
* Renal insufficiency
* Severe comorbidities requiring prompt management

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population who visited our center for gastric cancer screening using serum assays
Sampling Method: Non-Probability Sample
Enrollment: 1490 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Young Lee, MD, PhD, Principal Investigator — Department of Internal Medicine, Konkuk University School of Medicine
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Moon HW, Ahn YS, Song JH, Kim JH, Sung IK. A Prospective Study on the Detection of Gastric Neoplasms Using Pepsinogen and Gastrin-17 Levels. Gut Liver. 2025 Jul 15;19(4):548-558. doi: 10.5009/gnl240544. Epub 2025 Apr 11. PMID 40211909

RESULTS

PARTICIPANT FLOW:
Groups:
- No Gastric Neoplasm Group: Individuals without gastric neoplasms
- Gastric Neoplasm Group: Individuals with gastric neoplasms
Period: Overall Study
Arm/Group | No Gastric Neoplasm Group | Gastric Neoplasm Group
Started | 1346 | 144
Completed | 979 | 122
Not Completed | 367 | 22

BASELINE CHARACTERISTICS:
Groups:
- No Gastric Neoplasm: Individuals without gastric neoplasms
- Gastric Neoplasm: Individuals with gastric neoplasms
- Total: Total of all reporting groups
Arm/Group | No Gastric Neoplasm | Gastric Neoplasm | Total
Number analyzed (Participants) | 979 | 122 | 1101
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15.5) | 66.8 (10.1) | 53.0 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 451 | 42 | 493
  Male | 528 | 80 | 608
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 979 | 122 | 1101
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Status of H. pylori infection [Number; unit: Number of individuals]
  Current | 355 | 88 | 443
  Past | 303 | 32 | 334
  Naive | 321 | 2 | 323

OUTCOME MEASURES:

1. Primary Outcome: Significant Blood Test Findings Correlated With Gastric Neoplasms
Description: Serum pepsinogen I/II ratios indicating the presence gastric neoplasms (Minimum and maximum ratios were 0.2 and 19.1, respectively. Lower ratios indicate worse outcome.)
Time Frame: 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- No Gastric Neoplasm: Without gastric neoplasms (n=979)
- Gastric Neoplasm: With gastric neoplasms (n=122)
Arm/Group | No Gastric Neoplasm | Gastric Neoplasm
Number analyzed (Participants) | 979 | 122
score on a scale | 9.9 (3.9) | 6.5 (3.2)

2. Secondary Outcome: Test Findings Correlated With the Presence of Gastric Neoplasms
Description: Gastrin-17 levels measured by the GastroPanel tests on the day of other serologic tests including pepsinogen levels and Helicobacter pylori IgG titers
Time Frame: 15 months
Measure: Median (Full Range); unit: pmol/L
Arm/Group | No Gastric Neoplasm | Gastric Neoplasm
Number analyzed (Participants) | 979 | 122
pmol/L | 2.9 [0.4 to 30] | 11.8 [0.4 to 30]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded on the day of examination and on the day of follow-up visit at the outpatient clinic. Time Frame 1: On the day of upper gastrointestinal endoscopy and blood tests Time Frame 2: Up to 6 months
Description: Adverse events were defined as symptoms that disturbed daily activities by requiring management to subside the symptoms. Adverse events include perforation, bleeding, infection, cardiopulmonary events, etc.
Arm/Group | No Gastric Neoplasm Group | Gastric Neoplasm Group
All-Cause Mortality (participants affected / at risk) | 0/979 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/979 | 0/122
Other Adverse Events (participants affected / at risk) | 21/979 | 4/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Gastric Neoplasm Group (N=979) | Gastric Neoplasm Group (N=122)
Perforation, bleeding, infection, etc. (Gastrointestinal disorders) | 0 (0) | 0 (0) — Gastrointestinal perforation, bleeding, and infection which required treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Gastric Neoplasm Group (N=979) | Gastric Neoplasm Group (N=122)
Hypoxemia (Injury, poisoning and procedural complications) | 21 (21) | 4 (4) — SpO2 was monitored using a pulse oximetry for upper gastrointestinal endoscopy. Only mild hypoxemia (which did not require further management) was noticed during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT05883345/Prot_SAP_000.pdf